CLINICAL TRIAL: NCT03403738
Title: Bounce Back Now: A Low-Cost Intervention to Facilitate Post-Disaster Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH10764
Record Dates: First submitted 2017-12-08; First posted 2018-01-19 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: single (outcomes assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual Care (Active Comparator): usual care plus comprehensive resource list
  Interventions: Behavioral: enhanced usual care
- BBN (Experimental): Bounce Back Now intervention
  Interventions: Behavioral: Bounce Back Now

INTERVENTIONS:
Behavioral: Bounce Back Now — web/smartphone-based intervention for disaster victims
  Arms: BBN
Behavioral: enhanced usual care — enhanced usual care with list of resources
  Arms: Enhanced usual Care

SUMMARY:
Disaster survivors need freely accessible resources to self-monitor their emotional recovery and help them address mental health needs they may develop after a disaster. The investigators will evaluate a novel, scalable, and highly sustainable smartphone/web-based intervention that is designed to address post-disaster PTSD and depressed mood. The intervention, Bounce Back Now, will be tested in a study with 5,000 disaster survivors and will be accessible via any internet-connected device (e.g., laptop, tablet, smartphone).

DETAILED DESCRIPTION:
Globally, an average of 390 disasters, 100,000 related deaths, 260 million disaster victims, and $140 billion in economic damages were recorded per year between 2002-2012. The U.S. is one of the top 5 countries-with China, Philippines, India, and Indonesia-most frequently affected by disasters. The adverse mental health effects of disasters are extraordinary and costly. Up to 38% of distressed survivors presenting to shelters and assistance centers have stress-related and adjustment disorders. Most survivors who develop disaster-related mental health problems do not receive services. The 2013 report of the International Federation of Red Cross and Red Crescent Societies calls for technology-based solutions to heighten access to disaster assistance resources. With US cellphone and smartphone ownership now topping 90% and 60%, respectively, opportunities are tremendous to create cost-efficient, scalable solutions that increase capacity to address mental health needs in disaster-affected communities. The investigators propose highly innovative, time-sensitive research to examine the effectiveness of a widely accessible, technology-based disaster mental health intervention.

Mental health recovery trajectories are highly variable in disaster settings. 7,14 Most survivors recover without intervention and may need nothing more than a brief symptom tracking resource (i.e., watchful waiting). Some develop mental health needs (e.g., post-traumatic stress, depression) for which a brief self-help intervention may aid recovery. Some have chronic mental health problems (pre-existing or disaster related) that necessitate formal treatment. Others (e.g., serious mental illness) may require immediate assistance. The proposed intervention, Bounce Back Now (BBN), addresses each level of need using a web/smartphone-based approach that builds on the investigator's prior work. BBN consists of 3 key components: (1) a symptom and activity-tracking component that we piloted in emergency department settings, (2) a self-help intervention that was found to be efficacious in a recent RCT with families affected by a tornado outbreak, and (3) a resource component that principally connects survivors to the SAMHSA-administered Disaster Distress Helpline (DDH) when immediate assistance is needed (e.g., serious mental illness) or when local mental health treatment referrals are needed or preferred.

This study will leverage the mental health workforce to recruit 5,000 disaster survivors via partnerships with the American Red Cross (ARC) and Office of the Assistant Secretary for Preparedness and Response (ASPR). These partnerships allow cost-efficient testing of interventions, recruitment of individuals at high risk for developing disaster-related mental health problems, and collection of data at the level of triage to aid in prediction of mental health needs and coordination of care. Participants will be randomly assigned to receive BBN vs. enhanced usual care (i.e., EUC; usual care plus comprehensive resource list). BBN will be optimized for smartphones but accessible from any device with an internet connection.

ELIGIBILITY:
Inclusion Criteria:

1. individuals must be aged 18 years and older who were directly or indirectly affected by the disaster.
2. individual must be at least 18 years of age
3. have access to an internet-accessible device or computer, and
4. be English-speaking (i.e., all of the intervention content will be developed in the English language; it is cost-prohibitive to develop the system in multiple language in the testing phase)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1357 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist-Civilian version (PCL) | we will measure change from baseline and 3, 6, and 12-month post assessment
  20-item scale that assesses symptoms of DSM-defined PTSD.
Patient-Reported Outcomes Measurement Information System (PROMIS) | we will measure change from baseline and 3, 6, and 12-month post assessment
  8-item measure to assess symptoms of depression according to DSM-V criteria.
Behavioral Activation for Depression Scale | we will measure change from baseline and 3, 6, and 12-month post assessment
  25-item measure to assess avoidance behavior as well as pleasant and social activities. Each item is rated on a 7-point Likert scale ranging from 0 (not at all) to 6 (completely). To score the BADS, items from all scales other than the Activation scale are reverse-coded and then all items are summed. To score the subscales, no items are reverse-coded. This process allows high scores on the total scale and the subscales to be represented by the scale and subscale names. In other words, for the total scale, higher scores represent increased activation, while for the Social Impairment subscale, higher scores represent increased social impairment.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Sleep Disturbance Scale | we will measure change from baseline and 3, 6, and 12-month post assessment
  8-tem measure to assess sleep disturbance and sleep-related impairment. The 8-items are answered on a 5-point Likert scale ranging from 1 (not at all) to 5 (Very much). To find the total raw score for a short form with all questions answered, sum the values of the response to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40.
Kessler 6 | we will measure change from baseline and 3, 6, and 12-month post assessment
  6-item screening scale for probable serious mental illness (SMI)
The Alcohol Use Disorders Identification Test-Consumption questionnaire (AUDIT-C) | we will measure change from baseline and 3, 6, and 12-month post assessment
  3-item screen that identifies hazardous drinkers or individuals with active alcohol use disorders. The AUDIT-C is scored on a scale of 0-12.
  Each AUDIT-C question has 5 answer choices. Points allotted are: a = 0 points, b = 1 point, c = 2 points, d = 3 points, e = 4 points. In men, a score of 4 or more is considered positive, optimal for identifying hazardous drinking or active alcohol use disorders. In women, a score of 3 or more is considered positive (same as above). Generally, the higher the score, the more likely it is that the patient's drinking is affecting his or her safety.
Medical Outcomes Study (MOS-SS) Social Support Survey | we will measure change from baseline and 3, 6, and 12-month post assessment
  measures emotional, instrumental and appraisal support

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Ruggiero, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States